CLINICAL TRIAL: NCT04190940
Title: Functional Interaction of Thalamus, Basal Ganglia, and the Cerebellum in Visuomotor Adaptation
Brief Title: Interactions of Brain Regions in Visuomotor Adaptation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21483
Record Dates: First submitted 2019-11-17; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: High Intensity Focused Ultrasound; Deep Brain Stimulation
Keywords: Ultrasound; Thalamus; Cerebellum; Basal Ganglia; Deep Brain Stimulation; High Intensity Focused Ultrasound
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Focused Ultrasound (Experimental): Patients receiving high intensity focused ultrasound as a treatment will be asked to complete the behavioral task pre and post their treatment.
  Interventions: Behavioral: Behavioral Assessment
- Deep Brain Stimulation (Experimental): Patients receiving deep brain stimulation as a treatment will be asked to complete the behavioral task while their DBS electrode is "on" and "off".
  Interventions: Behavioral: Behavioral Assessment

INTERVENTIONS:
Behavioral: Behavioral Assessment — Patients will be asked to complete the behavioral assessment before and after their HIFU treatment or "on" and "off" their DBS treatment.

SUMMARY:
The purpose of this study is to better understand the roles the cerebellum, basal ganglia, and thalamus play in motor learning. Patients undergoing High Intensity Focused Ultrasound (HIFU) treatment will be receiving an ablation procedure to their thalamus as a part of their medical procedure. Participation in this study will include completing a behavioral task before and after the procedure to see how motor learning task performance differs with and without the thalamus. Similarly, patients undergoing Deep Brain Stimulation (DBS) treatment will have an electrode implanted in their thalamus as a part of their medical procedures. Participation in this study will include completing the motor learning task performance "on" and "off" thalamic electrical stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Be a patient receiving either high intensity focused ultrasound treatment or deep brain stimulation treatment for Tremor
* Able to provide informed consent and complete study procedures
* Must speak English
* Age 18-85

Exclusion Criteria:

* Not receiving one of the specified inclusion criteria
* Unable to provide consent or complete study procedures
* Women who self-report pregnancy
* Patients who are currently incarcerated

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2019-04-18 (Actual); Primary Completion 2021-04-17 (Estimated); Study Completion 2021-04-17 (Estimated)

PRIMARY OUTCOMES:
Performance Error on Visuomotor Task | baseline, a week after HIFU treatment, several weeks after DBS implantation
  The visuomotor task has practice, baseline, and experimental trials. Performance on the task will be compared between groups (HIFU treatment and DBS treatment) before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided